CLINICAL TRIAL: NCT06020560
Title: Cluster-randomized Trial of Low Molecular Weight Heparins - Directly Through EPIC
Brief Title: Study of Low Molecular Weight Heparins
Acronym: DANHEP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Kasper Iversen, Clinical Professor, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DANHEP
Record Dates: First submitted 2023-03-27; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Anticoagulant; Venous Thromboembolism; Prophylaxis; Treatment
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dalteparin (Active Comparator)
  Interventions: Drug: Tinzaparin profiled syringe
- Tinzaparin (Active Comparator)
  Interventions: Drug: Dalteparin Prefilled Syringe

INTERVENTIONS:
Drug: Dalteparin Prefilled Syringe — Patients will via a software module (Through a patient journal system) be allocated to either dalteparin or tinzaparin. Clusters are timeframes of 1 hour.
  Arms: Tinzaparin
Drug: Tinzaparin profiled syringe — Patients will via a software module (Through a patient journal system) be allocated to either dalteparin or tinzaparin. Clusters are timeframes of 1 hour.
  Arms: Dalteparin

SUMMARY:
DANHEP is a cluster randomized study of two different low molecular weight heparins. Parenteral anticoagulants are used in a variety of settings, including treatment and prevention of venous thromboembolism in cancer patients, medical patients, and surgical patients, along with the use as adjuvant therapy for coronary syndromes. The most frequently used parenteral anticoagulants in Denmark, include the two different low molecular weight heparins; dalteparin and tinzaparin. The two drugs are considered equally efficient and safe regarding treatment and prevention of thrombosis and risk of bleeding. Importantly, there is a lack of evidence regarding whether these drugs are in fact comparable. The aim of this study is therefore to investigate the comparative safety and efficacy of the two different low molecular weight heparins (dalteparin and tinzaparin using cluster randomization in patients with an indication for low molecular weight heparins.

ELIGIBILITY:
Inclusion Criteria:

* All patients with indication for low molecular weight heparin

Exclusion Criteria:

* Patients under the age of 18
* Patients who are incapable of understanding the written material received
* Patients who after being informed in writing chooses not to participate
* Patients with contraindications for low molecular weight heparins as described in the SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65000 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-03-23 (Estimated); Study Completion 2025-03-23 (Estimated)

PRIMARY OUTCOMES:
30-day all-cause mortality and bleeding requiring blood transfusion | 30 days
  To evaluate whether treatment with any of the low molecular weight heparins will increase the risk of bleeding requiring blood transfusion during admission or death within 30 days in patients with indication for low molecular weight heparins.

SECONDARY OUTCOMES:
30-day all-cause mortality | 30 days
  Risk of all-cause mortality within 30 days of administering one of the studied drugs
365-day all-cause mortality | 365 days
  Risk of all-cause mortality within 365 days of administering one of the studied drugs
Blood transfusion during admission | 90 days
  Blood transfusion defined from use of blood products
90 day risk of pulmonary embolism | 90 days
  Risk of pulmonary embolism within 90 days of administering one of the drugs studied
90 day risk of deep venous thrombosis | 90 days
  Risk of pulmonary embolism within 90 days of administering one of the drugs studied
Heparin induced thrombocytopenia | 90 days
  Risk of heparin induced thrombocytopenia defined by; thrombocytes less than 150 x 109/l and presence of HIT antibodies
Liver failure | 90 days
  Risk of liver failure defined by ALAT 3X upper limit of normal
Length of hospital admission | Admission time (up to 1 year from inclusion measured in days)
  Length of hospital admission
Days alive out of hospital | Time out of hospital (up to 1 year from inclusion measured in days)
  Days alive out of hospital

OTHER OUTCOMES:
Pregnancy loss | 9 months
  Risk of pregnancy loss during treatment with either of the two drugs studied
Stillbirth | 9 months
  Risk of stillbirth during treatment with either of the two drugs studied
Antepartum bleeding | 9 months
  Risk of antepartum bleeding during treatment with either of the two drugs studied
Postpartum bleeding | up to 365 days
  Risk of postpartum bleeding during treatment with either of the two drugs studied
Placental complications | 9 months
  Risk of placental complications (Abruptio placenta, placenta prevue) during treatment with either of the two drugs studied
Preeclampsia | 9 months
  Risk of preeclampsia and eclampsia during treatment with either of the two drugs studied

CONTACTS AND LOCATIONS:
Locations (9):
- Denmark (9):
  - Amager-Hvidovre Hospital, Copenhagen
  - Frederiksberg and Bispebjerg Hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - Herlev and Gentofte Hospital, Herlev
  - Nordsjællands Hospital, Hillerød
  - Nykøbing Falster Hospital, Nykøbing Falster
  - Næstved, Ringsted, Slagelse Hospital, Næstved
  - Roskilde, Køge Hospital, Roskilde
  - Bornholm Hospital, Rønne

IPD SHARING:
Plan to Share IPD: No